CLINICAL TRIAL: NCT03207867
Title: A Phase 2, Multi-center, Open Label Study of NIR178 in Combination With PDR001 in Patients With Selected Advanced Solid Tumors and Non-Hodgkin Lymphoma
Brief Title: A Phase 2 Study of NIR178 in Combination With PDR001 in Patients With Solid Tumors and Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIR178X2201; 2017-000241-49 (EudraCT Number)
Record Dates: First submitted 2017-06-19; First posted 2017-07-05 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: NSCLC, Non Small Cell Lung Cancer; RCC, Renal Cell Cancer; Pancreatic Cancer; Urothelial Cancer; Head and Neck Cancer; DLBCL, Diffused Large B Cell Lymphoma; MSS, Microsatellite Stable Colon Cancer; TNBC, Triple Negative Breast Cancer; Melanoma; mCRPC, Metastatic Castration Resistant Prostate Cancer
Keywords: Immunotherapy; A2aR; PDR001; NIR178; NSCLC; solid tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Pancreatic Neoplasms; Head and Neck Neoplasms; Spinocerebellar Degenerations; Triple Negative Breast Neoplasms; Melanoma | interventions — spartalizumab

STUDY DESIGN:
Intervention Model Description: Part 1, Part 3 and the Japanese safety run-in part were not randomized. In Part 2, patients were randomized to one of the 3 treatment arms in a ratio of 1:1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NIR178 + PDR001 (Experimental): Part 1: NIR178 continuously in combination with PDR001 400mg every 4 weeks. The part 1 enrolled 9 different tumor types.
  Interventions: Drug: NIR178; Drug: PDR001
- NIR178 BID Intermittent + PDR001 (Experimental): Part 2: Three different dosing schedules of NIR178 twice daily (BID) including continuous and two intermittent in combination with PDR001
  Interventions: Drug: NIR178; Drug: PDR001
- Part 3 (Experimental): Further evaluation of optimal intermittent or continuous schedule of NIR178 in combination with PDR001 (if selected based on results of Part 2). A film-coated tablet of NIR178 was assessed.
  Interventions: Drug: NIR178; Drug: PDR001
- Japanese safety run-in part (Experimental): Different dosing schedules of NIR178 were explored.
  Interventions: Drug: NIR178; Drug: PDR001

INTERVENTIONS:
Drug: NIR178 — NIR178, a new, non-xanthine based compound, is a potent oral adenosine A2a receptor against antagonist being developed by Novartis.
  NIR178 was administered orally twice daily (BID) as a capsule (Part 1, Part 2 and Japanese safety run-in) and as a film-coated table (Part 3). There were up to 3 dose levels assessed: 80, 160 and 240 mg. Three alternative dosing schedules were evaluated: continuous (Part 1, Part 2, Part 3, Japanese safety run-in), 2 weeks on/2 weeks off (Part 2) and 1 week on/1 week off (Part 2).
  Each cycle consisted of 28 days.
  Other Names: taminadenant
Drug: PDR001 — PDR001 is a human monoclonal antibody (MAb) administered on Day 1 of each cycle. PDR001 400 mg was administered via intravenous (i.v.) infusion over 30 minutes every 4 weeks (Q4W).
  Other Names: spartalizumab

SUMMARY:
The purpose of this phase 2 study is to evaluate the efficacy and safety of NIR178 in combination with PDR001 in multiple solid tumors and diffuse large B-cell lymphoma (DLBCL) and further explore schedule variations of NIR178 to optimize immune activation through inhibition of A2aR.

DETAILED DESCRIPTION:
This is an open-label multi-part, phase II study evaluating the combination of NIR178 and PDR001 in patients with advanced solid tumors and diffuse large B cell lymphoma (DLBCL).

The study has three parts:

* Part 1: Multi-arm Bayesian adaptive signal finding design in solid tumors and diffuse large B cell lymphoma (DLBCL) with continuous dosing of NIR178 in combination with PDR001.
* Part 2: Exploration of continuous and intermittent NIR178 schedules in combination with PDR001 in patients with advanced non-small cell lung cancer (NSCLC).
* Part 3: Further evaluation of optimal intermittent or continuous schedule of NIR178 in combination with PDR001 (if selected based on results of Part 2). As of protocol amendment 6, Part 3 explored the safety and pharmacokinetics of the film-coated tablet (FCT) formulation of NIR178 continuous dosing in combination with PDR001 in tiple negative breast cancer (TNBC) patients.

In addition, a separate safety run-in part was conducted in Japan in order to adequately characterize the safety and pharmacokinetic profiles of NIR178 as a single-agent and in combination with PDR001.

Patients enrolled in this study received NIR178 either twice daily (BID) continuously or based on the assigned intermittent schedule within 60 minutes prior to PDR001 infusion. PDR001 400 mg was administered via IV infusion over 30 minutes once every 4 weeks. Each treatment cycle was 28 days. Patients enrolled in the Japanese safety run-in part received NIR178 as single agent for the first cycle (28 days). If the patients completed Cycle 1 without experiencing dose limiting toxicities (DLTs), they initiated combination therapy with PDR001 starting Cycle 2 onwards, and continued at the same dose of NIR178. An additional cohort in the Japanese safety run-in part of the study received NIR178 in combination with PDR001 starting with Cycle 1. If the patients complete Cycle 1 without experiencing DLTs, they continued to receive combination treatment.

Patients received treatment with the combination until disease progression (assessed by investigator per immune-related response criteria (iRECIST) or Cheson 2014), unacceptable toxicity, death or discontinuation from study treatment for any other reason (e.g., withdrawal of consent, start of a new anti-neoplastic therapy or at the discretion of the investigator), otherwise known as End of Treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age. For Japan only: written consent is necessary both from the patient and his/her legal representative if he/she is under the age of 20 years.
* Histologically documented advanced or metastatic solid tumors or lymphomas Part 1: histologically confirmed renal cell carcinoma (RCC), pancreatic cancer, urothelial cancer, head and neck cancer, diffuse large B-cell lymphoma (DLBCL), microsatellite stable (MSS) colon cancer, triple negative breast cancer (TNBC), melanoma, metastatic castration resistant prostate cancer (mCRPC) Part 2: histologically confirmed diagnosis of advanced/metastatic NSCLC. For those with mixed histology, there must be a predominant histology Part 3: histologically confirmed diagnosis of selected advanced/metastatic malignancies. Part 3 will be opened to further assess TNBC patients with a PD-L1 SP-142 IC score of 0 (<1%). A second tumor group will be considered for Part 3 after completion of Part 1.
* Patient (except for those participating in Japanese safety run-in) must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Patient must be willing to undergo a new tumor biopsy at screening, and again during therapy on this study.
* Safety run-in part in Japanese patients can enroll any tumor type included in part 1, 2 and 3.

The collection of recent sample is permitted under the following conditions (both must be met):

Biopsy was collected ≤ 6 months before 1st dose of study treatment and available at the site.

No immunotherapy was given to the patient since collection of biopsy.

- Part 1 - 3 only: Patients (other than those with DLBCL) must previously have received at least 1 and no more than 3 prior lines of therapy for their disease (with the exception of IO-pretreated cutaneous melanoma, HNSCC and RCC), unless considered inappropriate for the patient (e.g. safety concern, label contraindication): Patients with NSCLC must have received a prior platinum-based combination. Patients with EGFR positive NSCLC with a T790M mutation must have progressed on osimertinib or discontinued due to toxicity.

Patients with head and neck cancer must have received a prior platinum-containing regimen.

Patients with bladder cancer must have received a prior platinum-containing regimen or be ineligible for cisplatin.

Patients with renal cell carcinoma must have received a prior VEGF tyrosine kinase inhibitor (TKI).

Patients with MSS colorectal cancer must have received (or be intolerant to) prior therapy with fluoropyrimidine-oxaliplatin- and irinotecan- based regimens.

Patients with triple negative breast cancer:. Part 1: must have received a prior taxane-containing regimen Part 3: should have received no more than 2 prior lines of therapy including taxane-based chemotherapy and should have a known PD-L1 status as per local available testing as determined by VENTANA PD-L1 SP142 Assay with IC score of 0 (<1%) Patients with DLBCL should be limited to those with no available therapies of proven clinical benefit Patients should have had prior autologous hematopoietic stem cell transplantation (auto-HSCT) or determined to be ineligible for auto-HSCT.

Patients with melanoma:

BRAF V600E wild type patients: must have received anti-PD-1/PD-L1 single agent, or in combination with anti-CTLA-4 therapy BRAF V600E mutant patients: must have received prior anti-PD-1/PD-L1 single-agent, or in combination with anti-CTLA-4 therapy. In addition, subjects must have received prior BRAF V600E inhibitor therapy, either single-agent or in combination with a MEK inhibitor

Patients with Metastatic Castration Resistant Prostate Cancer (mCRPC):

* Of the 1-3 prior lines of therapy, patients must have received and failed at least one line of treatment after emergence of castration resistant disease
* Patients must not have received prior immunotherapy (previous immune checkpoint inhibitors; single agent and/or combination therapy with anti-CTLA-4, anti-PD-1, anti-PD-L1), except for NSCLC patients enrolled in part 3 and Japanese safety run-in part.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral computer tomography (CT) scan, Magnetic Resonance Imaging (MRI), or calipers by clinical exam.

Exclusion Criteria:

* Ongoing or prior treatment with A2aR inhibitors. Patients previously treated with A2aR inhibitors for non-oncologic indications (e.g. Parkinson's disease) may be considered for enrollment on a case by case basis.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of PDR001, with the exception of intranasal/inhaled corticosteroids or systemic corticosteroids at physiological doses (not exceeding equivalent of 10 mg/day of prednisone)
* History of another primary malignancy except for:

Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of study drug and of low potential risk for recurrence Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease Adequately treated carcinoma in situ without evidence of disease

* Active or prior documented autoimmune disease within the past 2 years. Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* More than 3 prior lines of therapy except for Japanese safety run-in part.
* History of interstitial lung disease or non-infectious pneumonitis
* Systemic anti-cancer therapy within 2 weeks of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity, e.g. mitomycin C and nitrosoureas, 6 weeks is indicated as washout period. For patients receiving anticancer immunotherapies, 4 weeks is indicated as the washout period. GnRH therapy to maintain effective testosterone suppression levels is allowed for mCRPC patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (5):
  - University of California, Los Angeles, Santa Monica, California
  - H Lee Moffitt Cancer Center and Research Institute ., Tampa, Florida
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - MD Anderson Cancer Center/University of Texas, Houston, Texas
  - The University of Wisconsin, Madison, Wisconsin
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Novartis Investigative Site, Blacktown, New South Wales, Australia
- Novartis Investigative Site, Salzburg, Austria
- Novartis Investigative Site, Liège, Belgium
- Novartis Investigative Site, Brno, Czech Republic, Czechia
- Novartis Investigative Site, Marseille, France
- Germany (2):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Koto Ku, Tokyo, Japan
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Sankt Gallen, Switzerland
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 21 investigative sites in 15 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations had to be completed within 21 days prior to the first dose of treatment except for the radiological tumor assessment which had to be performed within 28 days prior to the first dose. After screening, the treatment period started on Cycle 1 Day 1.
Groups:
- Part 1: RCC naïve 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with renal cell carcinoma (RCC) who had not been previously treated with immuno-oncology therapy
- Part 1: RCC naïve 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with renal cell carcinoma (RCC) who had not been previously treated with immuno-oncology therapy
- Part 1: RCC Pre 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with renal cell carcinoma (RCC) who had been pretreated with immuno-oncology therapy
- Part 1: Pancreatic 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with pancreatic cancer
- Part 1: Urothelial 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with urothelial cancer
- Part 1: H-N naïve 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with squamous cell carcinoma of head and neck (HNSCC) who had not been previously treated with immuno-oncology therapy
- Part 1: H-N Pre 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with squamous cell carcinoma of head and neck (HNSCC) who had been pretreated with immuno-oncology therapy
- Part 1: H-N Pre 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with squamous cell carcinoma of head and neck (HNSCC) who had been pretreated with immuno-oncology therapy
- Part 1: MSS CRC wt 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with microsatellite stable colorectal cancer (MSS CRC) with RAS wildtype
- Part 1: MSS CRC mu 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with microsatellite stable colorectal cancer (MSS CRC) with RAS mutant
- Part 1: MSS CRC Unk 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with microsatellite stable colorectal cancer (MSS CRC) with unknown RAS status
- Part 1: TNBC 160 mg; Part 3: TNBC 160 mg Cont: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with triple negative breast cancer (TNBC)
- Part 1: Melanoma naïve 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with cutaneous melanoma who had not been previously treated with immuno-oncology therapy
- Part 1: Melanoma Pre 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with cutaneous melanoma who had been pretreated with immuno-oncology therapy
- Part 1: DLBCL 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with diffuse large B-cell lymphoma (DLBCL)
- Part 1: DLBCL 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with diffuse large B-cell lymphoma (DLBCL)
- Part 1: mCRPC 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with metastatic castration resistant prostate cancer (mCRPC)
- Part 2: NSCLC 160 mg Cont: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with non-small cell lung cancer (NSCLC)
- Part 2: NSCLC 160 mg 2wk-on/2wk-off: NIR178 160 mg twice daily 2 weeks on/2 weeks off in combination with PDR001 in patients with non-small cell lung cancer (NSCLC)
- Part 2: NSCLC 160 mg 1wk-on/1wk-off: NIR178 160 mg twice daily 1 week on/1 week off in combination with PDR001 in patients with non-small cell lung cancer (NSCLC)
- JSR: 80 mg Cont: NIR178 80 mg twice daily continuous in combination with PDR001 (starting Cycle 2 Day 1) in the Japan safety run-in
- JSR: 160 mg Cont: NIR178 160 mg twice daily continuous in combination with PDR001 (starting Cycle 2 Day 1) in the Japan safety run-in
- JSR: 240 mg Cont: NIR178 140 mg twice daily continuous in combination with PDR001 (starting Cycle 1 Day 1) in the Japan safety run-in
Period: Overall Study
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: MSS CRC Unk 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Started | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 12 | 27 | 29 | 2 | 30 | 3 | 13 | 13 | 6 | 15 | 22 | 20 | 20 | 6 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 12 | 27 | 29 | 2 | 30 | 3 | 13 | 13 | 6 | 15 | 22 | 20 | 20 | 6 | 3 | 3 | 3
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 5 | 0 | 3 | 2 | 0 | 0 | 0 | 4 | 2 | 0 | 4 | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 7 | 7 | 9 | 10 | 11 | 10 | 9 | 8 | 19 | 23 | 2 | 24 | 3 | 11 | 9 | 5 | 10 | 14 | 13 | 14 | 6 | 3 | 3 | 3
Not completed — Patient/guardian Decision | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 3 | 4 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: MSS CRC Unk 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont | Total
Number analyzed (Participants) | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 12 | 27 | 29 | 2 | 30 | 3 | 13 | 13 | 6 | 15 | 22 | 20 | 20 | 6 | 3 | 3 | 3 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.86) | 60.0 (11.96) | 60.6 (8.54) | 60.4 (8.98) | 66.9 (9.63) | 61.6 (7.13) | 59.4 (9.05) | 60.2 (7.07) | 56.5 (9.04) | 58.1 (11.21) | 46.0 (15.56) | 49.8 (10.81) | 50.3 (20.65) | 54.2 (14.87) | 55.0 (18.65) | 61.5 (13.10) | 68.3 (8.14) | 65.0 (9.02) | 61.8 (9.51) | 64.2 (8.94) | 58.5 (16.16) | 61.3 (10.69) | 57.0 (9.54) | 44.3 (8.33) | 59.5 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 6 | 5 | 2 | 3 | 3 | 9 | 8 | 1 | 30 | 1 | 3 | 7 | 3 | 0 | 7 | 7 | 8 | 6 | 3 | 1 | 1 | 119
  Male | 8 | 12 | 9 | 8 | 9 | 13 | 8 | 9 | 18 | 21 | 1 | 0 | 2 | 10 | 6 | 3 | 15 | 15 | 13 | 12 | 0 | 0 | 2 | 2 | 196
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 3 | 10 | 13 | 5 | 14 | 9 | 12 | 20 | 23 | 2 | 21 | 1 | 13 | 7 | 0 | 13 | 10 | 7 | 7 | 1 | 0 | 0 | 0 | 200
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 10
  Asian | 2 | 8 | 0 | 0 | 8 | 1 | 0 | 0 | 6 | 1 | 0 | 2 | 2 | 0 | 4 | 6 | 2 | 11 | 13 | 12 | 0 | 0 | 0 | 0 | 78
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 5
  Unknown | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 7 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 21

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Overall Response Rate (ORR) Per RECIST v1.1 for Solid Tumors
Description: ORR is the percentage of patients with a best overall response of complete response (CR) or partial response (PR), based on local investigator assessment per Response Evaluation Criteria for Solid Tumors (RECIST) v1.1.
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 3.9 years
Population: All patients from Part 1 who received at least 1 full or partial dose of assigned combination of study drugs and were included in the selected advanced solid tumors groups defined in the study protocol for efficacy assessment: RCC naïve 160 mg, RCC naïve 240 mg, RCC pre 240 mg, pancreatic 160 mg, urothelial 160 mg, H-N naïve 160 mg, H-N pre 160 mg, MSS CRC wt 160 mg, MSS CRC mu 160 mg, TNBC 160 mg, melanoma pre 160 mg and mCRPC 240 mg
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 27 | 29 | 30 | 13 | 15
percentage of participants | 27.3 [7.9 to 56.4] | 25.0 [7.2 to 52.7] | 0 [0.0 to 23.8] | 0 [0.0 to 19.3] | 7.1 [0.4 to 29.7] | 13.3 [2.4 to 36.3] | 0 [0.0 to 23.8] | 0 [0.0 to 10.5] | 3.4 [0.2 to 15.3] | 10.0 [2.8 to 23.9] | 0 [0.0 to 20.6] | 0 [0.0 to 18.1]

2. Primary Outcome: Part 1: Overall Response Rate (ORR) Per Cheson 2014 for DLBCL
Description: ORR is the percentage of patients with a best overall response of complete response (CR) or partial response (PR), based on local investigator assessment per Cheson 2014 criteria for diffuse large B-cell lymphoma (DLBCL).
  For Cheson 2014 criteria, CR= Target nodes/nodal masses must regress to ≤1.5 cm in longest diameter (LDi), no extralymphatic sites of disease, absent non-measured lesions, organ enlargement regress to normal, no new lesions, and bone marrow normal by morphology (if indeterminate, immunohistochemistry negative); PR= ≥50% decrease in the sum of the product of the perpendicular diameters (SPD) of up to 6 target measurable nodes, absent or regressed non-measured lesions, spleen must have regressed by >50% in length beyond normal, and no new lesions.
Time Frame: Up to 2.5 years
Population: All patients from Part 1 who received at least 1 full or partial dose of assigned combination of study drugs and were included in the selected lymphoma group defined in the study protocol for efficacy assessment: DLBCL 160 mg
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: DLBCL 160 mg
Number analyzed (Participants) | 13
percentage of participants | 15.4 [2.8 to 41.0]

3. Primary Outcome: Part 2: Overall Response Rate (ORR) Per RECIST v1.1 for Solid Tumors
Description: ORR is the percentage of patients with a best overall response of complete response (CR) or partial response (PR), based on local investigator assessment per RECIST v1.1.
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 4.7 years
Population: All patients from Part 2 who were randomized to the study treatment dosing schedule.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 22 | 20 | 20
percentage of participants | 9.1 [1.6 to 25.9] | 0 [0.0 to 13.9] | 10.0 [1.8 to 28.3]

4. Primary Outcome: Part 3: Overall Response Rate (ORR) Per RECIST v1.1 for Solid Tumors
Description: as for outcome 3
Time Frame: Up to 0.5 years
Population: All patients from Part 3 who received at least 1 full or partial dose of assigned combination of study drugs.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 6
percentage of participants | 16.7 [0.9 to 58.2]

5. Secondary Outcome: Part 1: Overall Response Rate (ORR) Per iRECIST for Solid Tumors
Description: ORR is the percentage of patients with a best overall response of complete response (iCR) or partial response (iPR), based on local investigator assessment per immune-related RECIST (iRECIST).
Time Frame: Up to 3.9 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 27 | 29 | 30 | 13 | 15
percentage of participants | 36.4 [13.5 to 65.0] | 25.0 [7.2 to 52.7] | 0 [0.0 to 23.8] | 0 [0.0 to 19.3] | 7.1 [0.4 to 29.7] | 13.3 [2.4 to 36.3] | 0 [0.0 to 23.8] | 0 [0.0 to 10.5] | 3.4 [0.2 to 15.3] | 10.0 [2.8 to 23.9] | 0 [0.0 to 20.6] | 0 [0.0 to 18.1]

6. Secondary Outcome: Part 2: Overall Response Rate (ORR) Per iRECIST for Solid Tumors
Description: as for outcome 5
Time Frame: Up to 4.7 years
Population: All patients from Part 2 who were randomized to the study treatment dosing schedule.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 22 | 20 | 20
percentage of participants | 9.1 [1.6 to 25.9] | 5.0 [0.3 to 21.6] | 15.0 [4.2 to 34.4]

7. Secondary Outcome: Part 3: Overall Response Rate (ORR) Per iRECIST for Solid Tumors
Description: as for outcome 5
Time Frame: Up to 0.5 years
Population: All patients from Part 3 who received at least 1 full or partial dose of assigned combination of study drugs.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 6
percentage of participants | 16.7 [0.9 to 58.2]

8. Secondary Outcome: Part 1: Mean Percentage Change in PSA From Baseline
Description: Prostate-specific antigen (PSA) levels were assessed in serum. Rising PSA is generally a manifestation of progression of prostate cancer.
Time Frame: Baseline, up to 0.8 years
Population: All patients from Part 1 who received at least 1 full or partial dose of assigned combination of study drugs and were included in the prostate cancer group defined in the study protocol for efficacy assessment: mCRPC 240 mg
Measure: Mean (Standard Deviation); unit: percentage change in PSA from baseline
Arm/Group | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 15
percentage change in PSA from baseline | 214.46 (329.459)

9. Secondary Outcome: Part 1: Disease Control Rate (DCR) Per RECIST v1.1 for Solid Tumors
Description: DCR is the percentage of patients with a best overall response of complete response (CR), partial response (PR), stable disease (SD) or Non-CR or Non-progressive disease (NCRNPD), based on local investigator assessment per Response Evaluation Criteria for Solid Tumors (RECIST) v1.1.
Time Frame: Up to 3.9 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 27 | 29 | 30 | 13 | 15
percentage of participants | 54.5 [27.1 to 80.0] | 66.7 [39.1 to 87.7] | 18.2 [3.3 to 47.0] | 0 [0.0 to 19.3] | 28.6 [10.4 to 54.0] | 40.0 [19.1 to 64.0] | 63.6 [35.0 to 86.5] | 25.9 [12.9 to 43.2] | 17.2 [7.0 to 32.9] | 33.3 [19.3 to 49.9] | 0 [0.0 to 20.6] | 46.7 [24.4 to 70.0]

10. Secondary Outcome: Part 1: Disease Control Rate (DCR) Per iRECIST for Solid Tumors
Description: DCR is the percentage of patients with a best overall response of complete response (iCR), partial response (iPR), stable disease (iSD) or Non-iCR or Non-unconfirmed progressive disease (NON-iCR or NON-iUPD), based on local investigator assessment per immune-related RECIST (iRECIST).
Time Frame: Up to 3.9 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 27 | 29 | 30 | 13 | 15
percentage of participants | 63.6 [35.0 to 86.5] | 66.7 [39.1 to 87.7] | 18.2 [3.3 to 47.0] | 0 [0.0 to 19.3] | 35.7 [15.3 to 61.0] | 40.0 [19.1 to 64.0] | 54.5 [27.1 to 80.0] | 25.9 [12.9 to 43.2] | 13.8 [4.9 to 28.8] | 36.7 [22.1 to 53.3] | 0 [0.0 to 20.6] | 46.7 [24.4 to 70.0]

11. Secondary Outcome: Part 1: Disease Control Rate (DCR) Per Cheson 2014 for DLBCL
Description: DCR is the percentage of patients with a best overall response of complete response (CR), partial response (PR) or stable disease (SD), based on local investigator assessment per Cheson 2014 criteria for diffuse large B-cell lymphoma (DLBCL).
Time Frame: Up to 2.5 years
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: DLBCL 160 mg
Number analyzed (Participants) | 13
percentage of participants | 23.1 [6.6 to 49.5]

12. Secondary Outcome: Part 2: Disease Control Rate (DCR) Per RECIST v1.1 for Solid Tumors
Description: as for outcome 9
Time Frame: Up to 4.7 years
Population: All patients from Part 2 who were randomized to the study treatment dosing schedule.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 22 | 20 | 20
percentage of participants | 36.4 [19.6 to 56.1] | 40.0 [21.7 to 60.6] | 35.0 [17.7 to 55.8]

13. Secondary Outcome: Part 2: Disease Control Rate (DCR) Per iRECIST for Solid Tumors
Description: as for outcome 10
Time Frame: Up to 4.7 years
Population: All patients from Part 2 who were randomized to the study treatment dosing schedule.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 22 | 20 | 20
percentage of participants | 36.4 [19.6 to 56.1] | 45.0 [25.9 to 65.3] | 45.0 [25.9 to 65.3]

14. Secondary Outcome: Part 3: Disease Control Rate (DCR) Per RECIST v1.1 for Solid Tumors
Description: as for outcome 9
Time Frame: Up to 0.5 years
Population: All patients from Part 3 who received at least 1 full or partial dose of assigned combination of study drugs.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 6
percentage of participants | 16.7 [0.9 to 58.2]

15. Secondary Outcome: Part 3: Disease Control Rate (DCR) Per iRECIST for Solid Tumors
Description: as for outcome 10
Time Frame: Up to 0.5 years
Population: All patients from Part 3 who received at least 1 full or partial dose of assigned combination of study drugs.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 6
percentage of participants | 16.7 [0.9 to 58.2]

16. Secondary Outcome: Part 1: Duration Of Response (DOR) Per RECIST v1.1 for Solid Tumors
Description: DOR only applies to patients for whom best overall response is complete response (CR) or partial response (PR) based on local investigator assessment per RECIST v1.1. DOR is defined as the time from the date of first documented response (CR or PR) to the date of first documented progression or death due to underlying cancer. If a patient did not have an event, DOR was censored at the date of last adequate tumor assessment.
  DOR was analyzed using Kaplan-Meier estimates as defined in the statistical analysis plan.
Time Frame: Up to 3.9 years
Population: All patients from Part 1 for whom best overall response was CR or PR and were included in the selected advanced solid tumors groups defined in the study protocol for efficacy assessment: RCC naïve 160 mg, RCC naïve 240 mg, RCC pre 240 mg, pancreatic 160 mg, urothelial 160 mg, H-N naïve 160 mg, H-N pre 160 mg, MSS CRC wt 160 mg, MSS CRC mu 160 mg, TNBC 160 mg, melanoma pre 160 mg and mCRPC 240 mg
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 3 | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 0 | 0
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events |  |

17. Secondary Outcome: Part 1: Duration Of Response (DOR) Per iRECIST for Solid Tumors
Description: DOR only applies to patients for whom best overall response is complete response (iCR) or partial response (iPR) based on local investigator assessment per iRECIST. DOR is defined as the time from the date of first documented response (iCR or iPR) to the date of first documented progression or death due to underlying cancer. If a patient did not have an event, DOR was censored at the date of last adequate tumor assessment.
  DOR was analyzed using Kaplan-Meier estimates as defined in the statistical analysis plan.
Time Frame: Up to 3.9 years
Population: All patients from Part 1 for whom best overall response was iCR or iPR and were included in the selected advanced solid tumors groups defined in the study protocol for efficacy assessment: RCC naïve 160 mg, RCC naïve 240 mg, RCC pre 240 mg, pancreatic 160 mg, urothelial 160 mg, H-N naïve 160 mg, H-N pre 160 mg, MSS CRC wt 160 mg, MSS CRC mu 160 mg, TNBC 160 mg, melanoma pre 160 mg and mCRPC 240 mg
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 4 | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 0 | 0
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events |  |

18. Secondary Outcome: Part 1: Duration Of Response (DOR) Per Cheson 2014 for DLBCL
Description: DOR only applies to patients for whom best overall response is complete response (CR) or partial response (PR) based on local investigator assessment per Cheson 2014 criteria for DLBCL. DOR is defined as the time from the date of first documented response (CR or PR) to the date of first documented progression or death due to underlying cancer. If a patient did not have an event, DOR was censored at the date of last adequate tumor assessment. DOR was analyzed using Kaplan-Meier estimates as defined in the statistical analysis plan.
Time Frame: Up to 2.5 years
Population: All patients from Part 1 for whom best overall response was CR or PR and were included in the selected lymphoma group defined in the study protocol for efficacy assessment: DLBCL 160 mg
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1: DLBCL 160 mg
Number analyzed (Participants) | 2
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events

19. Secondary Outcome: Part 2: Duration Of Response (DOR) Per RECIST v1.1 for Solid Tumors
Description: as for outcome 16
Time Frame: Up to 4.7 years
Population: All patients from Part 2 for whom best overall response was CR or PR
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 2 | 0 | 2
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events

20. Secondary Outcome: Part 2: Duration Of Response (DOR) Per iRECIST for Solid Tumors
Description: as for outcome 17
Time Frame: Up to 4.7 years
Population: All patients from Part 2 for whom best overall response was iCR or iPR
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 2 | 1 | 3
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events

21. Secondary Outcome: Part 3: Duration Of Response (DOR) Per RECIST v1.1 for Solid Tumors
Description: as for outcome 16
Time Frame: Up to 0.5 years
Population: All patients from Part 3 for whom best overall response was CR or PR
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 1
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events

22. Secondary Outcome: Part 3: Duration Of Response (DOR) Per iRECIST for Solid Tumors
Description: as for outcome 17
Time Frame: Up to 0.5 years
Population: All patients from Part 3 for whom best overall response was iCR or iPR
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 1
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events

23. Secondary Outcome: Part 1: Progression-Free Survival (PFS) Per RECIST v1.1 for Solid Tumors
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause, whichever happened first. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on local investigator assessment per RECIST v1.1.
  PFS was analyzed using Kaplan-Meier estimates as defined in the statistical analysis plan.
Time Frame: Up to 3.9 years
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 27 | 29 | 30 | 13 | 15
months | 3.5 [1.9 to 15.4] | 7.2 [1.8 to 8.6] | 1.9 [1.7 to 2.0] | 1.7 [1.6 to 1.7] | 1.9 [1.7 to 3.5] | 2.0 [1.6 to 3.7] | 3.5 [1.7 to 3.7] | 1.7 [1.6 to 1.9] | 1.9 [1.7 to 2.0] | 1.7 [1.6 to 1.9] | 1.8 [1.6 to 1.9] | 3.7 [1.7 to 5.3]

24. Secondary Outcome: Part 1: Progression-Free Survival (PFS) Per iRECIST for Solid Tumors
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause, whichever happened first. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on local investigator assessment per iRECIST.
  PFS was analyzed using Kaplan-Meier estimates as defined in the statistical analysis plan.
Time Frame: Up to 3.9 years
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 27 | 29 | 30 | 13 | 15
months | 8.7 [2.1 to NA] — Not estimable due to insufficient number of participants with events | 7.2 [1.8 to NA] — Not estimable due to insufficient number of participants with events | 1.9 [1.7 to 2.0] | 1.7 [1.1 to 1.7] | 2.1 [1.7 to 3.5] | 2.0 [1.6 to 3.7] | 3.5 [1.7 to 3.7] | 1.8 [1.6 to 2.0] | 1.9 [1.7 to 2.0] | 1.8 [1.6 to 3.5] | 1.8 [1.6 to 1.9] | 3.7 [1.7 to 5.3]

25. Secondary Outcome: Part 1: Progression-Free Survival (PFS) Per Cheson 2014 for DLBCL
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause, whichever happened first. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on local investigator assessment per Cheson 2014 for DLBCL.
  PFS was analyzed using Kaplan-Meier estimates as defined in the statistical analysis plan.
Time Frame: Up to 2.5 years
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1: DLBCL 160 mg
Number analyzed (Participants) | 13
months | 1.7 [1.4 to 2.2]

26. Secondary Outcome: Part 2: Progression-Free Survival (PFS) Per RECIST v1.1 for Solid Tumors
Description: as for outcome 23
Time Frame: Up to 4.7 years
Population: All patients from Part 2 who were randomized to the study treatment dosing schedule.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 22 | 20 | 20
months | 2.0 [1.8 to 3.8] | 2.1 [1.7 to 3.7] | 1.9 [1.7 to 3.7]

27. Secondary Outcome: Part 2: Progression-Free Survival (PFS) Per iRECIST for Solid Tumors
Description: as for outcome 24
Time Frame: Up to 4.7 years
Population: All patients from Part 2 who were randomized to the study treatment dosing schedule.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 22 | 20 | 20
months | 2.1 [1.8 to 3.8] | 2.2 [1.8 to 3.7] | 2.8 [1.7 to 9.0]

28. Secondary Outcome: Part 3: Progression-Free Survival (PFS) Per RECIST v1.1 for Solid Tumors
Description: as for outcome 23
Time Frame: Up to 0.5 years
Population: All patients from Part 3 who received at least 1 full or partial dose of assigned combination of study drugs.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 6
months | 1.6 [0.9 to 1.8]

29. Secondary Outcome: Part 3: Progression-Free Survival (PFS) Per iRECIST for Solid Tumors
Description: as for outcome 24
Time Frame: Up to 0.5 years
Population: All patients from Part 3 who received at least 1 full or partial dose of assigned combination of study drugs.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 6
months | 1.6 [0.9 to 1.8]

30. Secondary Outcome: Part 1: 2-year Overall Survival (OS)
Description: OS represents the percentage of participants who are alive after the start of study treatment. OS at 2 years was estimated using the Kaplan-Meier method as defined in the statistical analysis plan (SAP).
Time Frame: 2 years
Population: All patients from Part 1 who received at least 1 full or partial dose of assigned combination of study drugs and were included in the selected cancer groups defined in the protocol for efficacy assessment: RCC naïve 160 mg, RCC naïve 240 mg, RCC pre 240 mg, pancreatic 160 mg, urothelial 160 mg, H-N naïve 160 mg, H-N pre 160 mg, MSS CRC wt 160 mg, MSS CRC mu 160 mg, TNBC 160 mg, melanoma pre 160 mg, DLBCL 160 mg and mCRPC 240 mg
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 11 | 12 | 11 | 14 | 14 | 15 | 11 | 27 | 29 | 30 | 13 | 13 | 15
percentage of participants | 63.6 [35.5 to 82.1] | 42.1 [14.6 to 67.8] | 27.3 [8.9 to 49.8] | NA [NA to NA] — Not estimable due to insufficient number of participants with events | 36.1 [15.0 to 57.9] | 33.3 [15.0 to 52.9] | 15.3 [1.9 to 41.2] | 22.1 [9.4 to 38.2] | 14.3 [4.3 to 29.9] | 30.8 [16.0 to 46.9] | NA [NA to NA] — Not estimable due to insufficient number of participants with events | 23.1 [7.5 to 43.6] | 31.4 [10.8 to 54.7]

31. Secondary Outcome: Part 2: 2-year Overall Survival (OS)
Description: OS represents the percentage of participants who are alive after the start of study treatment. OS at 2 years was estimated using the Kaplan-Meier method as defined in the statistical analysis plan.
Time Frame: 2 years
Population: All patients from Part 2 who were randomized to the study treatment dosing schedule.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 22 | 20 | 20
percentage of participants | 33.6 [15.5 to 52.9] | 22.7 [7.5 to 42.7] | 39.7 [20.3 to 58.6]

32. Secondary Outcome: Part 3: 2-year Overall Survival (OS)
Description: as for outcome 31
Time Frame: 2 years
Population: All patients from Part 3 who received at least 1 full or partial dose of assigned combination of study drugs.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 6
percentage of participants | NA [NA to NA] — Not estimable due to insufficient number of participants with events

33. Secondary Outcome: Part 1: Change From Baseline in CD8 Percent Marker Area in Tumor Tissue
Description: The tumor expression of CD8 was measured by immunohistochemical (IHC) methods. Newly obtained pre- and on-treatment paired tumor samples were required and collected at screening and after approximately two cycles of therapy.
Time Frame: Screening and on-treatment (Cycle 2 Day 1 or Day 15). The duration of one cycle was 28 days.
Population: All patients from Part 1 who received any study drug, had paired tumor samples, had a valid assessment for the outcome measure and were included in the selected cancer groups defined in the protocol for efficacy assessment: RCC naïve 160 mg, RCC naïve 240 mg, RCC pre 240 mg, pancreatic 160 mg, urothelial 160 mg, H-N naïve 160 mg, H-N pre 160 mg, MSS CRC wt 160 mg, MSS CRC mu 160 mg, TNBC 160 mg, melanoma pre 160 mg, DLBCL 160 mg and mCRPC 240 mg
Measure: Mean (Standard Deviation); unit: CD8 percent marker area
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve 240 mg | Part 1: RCC Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve 160 mg | Part 1: H-N Pre 160 mg | Part 1: MSS CRC wt 160 mg | Part 1: MSS CRC mu 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: mCRPC 240 mg
Number analyzed (Participants) | 2 | 5 | 3 | 2 | 6 | 5 | 4 | 7 | 9 | 10 | 4 | 1 | 4
CD8 percent marker area | 10.93 (14.227) | 10.53 (12.456) | 0.70 (2.645) | -0.81 (0.537) | 0.96 (1.345) | 1.63 (2.372) | -0.42 (1.477) | 0.70 (1.141) | -0.01 (1.164) | 4.86 (3.751) | 0.16 (0.540) | 7.84 | 2.67 (4.156)

34. Secondary Outcome: Part 2: Change From Baseline in CD8 Percent Marker Area in Tumor Tissue
Description: as for outcome 33
Time Frame: Screening and on-treatment (Cycle 2 Day 1 or Day 15). The duration of one cycle was 28 days.
Population: All patients from Part 2 who received any study drug, had paired tumor samples and had a valid assessment for the outcome measure
Measure: Mean (Standard Deviation); unit: CD8 percent marker area
Arm/Group | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off
Number analyzed (Participants) | 6 | 4 | 4
CD8 percent marker area | 3.81 (4.551) | -2.35 (5.586) | 1.23 (2.955)

35. Secondary Outcome: Part 3: Change From Baseline in CD8 Percent Marker Area in Tumor Tissue
Description: as for outcome 33
Time Frame: Screening and on-treatment (Cycle 2 Day 1 or Day 15). The duration of one cycle was 28 days.
Population: All patients from Part 3 who received any study drug, had paired tumor samples and had a valid assessment for the outcome measure
Measure: Mean (Standard Deviation); unit: CD8 percent marker area
Arm/Group | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 1
CD8 percent marker area | 0.26

36. Secondary Outcome: Part 1, 2 and 3: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: Number of participants with AEs (any AE regardless of seriousness) and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
  The on-treatment period is defined from the day of first administration of study treatment up to 30 days after the date of its last administration.
Time Frame: Up to 4 years (Part 1), 4.8 years (Part 2) and 0.6 years (Part 3)
Population: All patients from Part 1, 2 and 3 who received at least 1 dose of NIR178 or PDR001. For the safety endpoints, patients at each study part with the same type of cancer who are treated at the same dose level and dosing schedule are pooled together, independently of the immune-oncology (IO) pretreatment status and RAS mutation status.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: RCC naïve + Pre 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with renal cell carcinoma (RCC), naïve and pretreated with immuno-oncology therapy
- Part 1: H-N naïve + Pre 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with squamous cell carcinoma of head and neck (HNSCC), naïve and pretreated with immuno-oncology therapy
- Part 1: MSS CRC 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with microsatellite stable colorectal cancer (MSS CRC) and RAS wildtype, RAS mutant and RAS unknown status
- Part 1: Melanoma naïve + Pre 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with cutaneous melanoma, naïve and pretreated with immuno-oncology therapy
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve + Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve + Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve + Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 11 | 23 | 14 | 14 | 26 | 12 | 58 | 30 | 16 | 13 | 6 | 15 | 22 | 20 | 20 | 6
Participants
  AEs | 10 | 22 | 14 | 14 | 26 | 12 | 57 | 29 | 15 | 13 | 5 | 14 | 22 | 18 | 18 | 6
  Treatment-related AEs | 7 | 16 | 9 | 9 | 16 | 9 | 34 | 23 | 6 | 11 | 2 | 12 | 15 | 14 | 9 | 4
  SAEs | 3 | 7 | 9 | 7 | 15 | 5 | 28 | 11 | 3 | 6 | 0 | 4 | 11 | 7 | 7 | 3
  Treatment-related SAEs | 0 | 2 | 2 | 1 | 3 | 2 | 7 | 2 | 0 | 2 | 0 | 2 | 6 | 3 | 0 | 0
  Fatal SAEs | 1 | 0 | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
  Treatment-related fatal SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

37. Secondary Outcome: Part 1, 2 and 3: Number of Participants With Dose Reductions and Dose Interruptions of NIR178
Description: Number of participants with at least one dose reduction of NIR178 and number of participants with at least one dose interruption of NIR178. Dose or schedule adjustments were permitted for patients who did not tolerate the protocol-specified dosing schedule.
Time Frame: Up to 3.9 years (Part 1), 4.7 years (Part 2) and 0.5 years (Part 3)
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve + Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve + Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve + Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 11 | 23 | 14 | 14 | 26 | 12 | 58 | 30 | 16 | 13 | 6 | 15 | 22 | 20 | 20 | 6
Participants
  At least one dose reduction | 2 | 1 | 0 | 2 | 8 | 1 | 7 | 3 | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 0
  At least one dose interruption | 6 | 9 | 2 | 8 | 12 | 3 | 20 | 9 | 3 | 3 | 1 | 5 | 8 | 5 | 4 | 0

38. Secondary Outcome: Part 1, 2 and 3: Number of Participants With Dose Reductions and Dose Interruptions of PDR001
Description: Number of participants with at least one dose reduction of PDR001 and number of participants with at least one dose interruption of PDR001. Dose or schedule adjustments were permitted for patients who did not tolerate the protocol-specified dosing schedule. Dose reductions were not permitted for PDR001.
Time Frame: Up to 3.9 years (Part 1), 4.7 years (Part 2) and 0.5 years (Part 3)
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve + Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve + Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve + Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 11 | 23 | 14 | 14 | 26 | 12 | 58 | 30 | 16 | 13 | 6 | 15 | 22 | 20 | 20 | 6
Participants
  At least one dose reduction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least one dose interruption | 6 | 7 | 1 | 6 | 9 | 1 | 13 | 8 | 2 | 0 | 0 | 2 | 6 | 4 | 2 | 0

39. Secondary Outcome: Part 1, 2 and 3: Dose Intensity of NIR178
Description: Dose intensity of NIR178 was calculated as cumulative actual dose in milligrams divided by duration of exposure in days.
Time Frame: Up to 3.9 years (Part 1), 4.7 years (Part 2) and 0.5 years (Part 3)
Population: as for outcome 36
Measure: Median (Full Range); unit: mg/day
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve + Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve + Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve + Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 11 | 23 | 14 | 14 | 26 | 12 | 58 | 30 | 16 | 13 | 6 | 15 | 22 | 20 | 20 | 6
mg/day | 316.7 [187 to 320] | 477.3 [321 to 480] | 320.0 [241 to 320] | 295.7 [140 to 320] | 309.8 [141 to 320] | 480.0 [272 to 480] | 320.0 [134 to 320] | 320.0 [179 to 320] | 320.0 [208 to 320] | 320.0 [233 to 320] | 480.0 [363 to 480] | 480.0 [382 to 496] | 320.0 [137 to 320] | 160.0 [96 to 173] | 160.0 [71 to 189] | 320.0 [319 to 320]

40. Secondary Outcome: Part 1, 2 and 3: Dose Intensity of PDR001
Description: Dose intensity of PDR001 was calculated as cumulative actual dose in milligrams divided by duration of exposure in days and then multiplied by 28 days.
Time Frame: Up to 3.9 years (Part 1), 4.7 years (Part 2) and 0.5 years (Part 3)
Population: as for outcome 36
Measure: Median (Full Range); unit: mg/28 days
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve + Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve + Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve + Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 11 | 23 | 14 | 14 | 26 | 12 | 58 | 30 | 16 | 13 | 6 | 15 | 22 | 20 | 20 | 6
mg/28 days | 394.2 [300 to 400] | 396.2 [267 to 431] | 400.0 [395 to 400] | 393.1 [350 to 400] | 398.2 [319 to 402] | 400.0 [365 to 407] | 400.0 [236 to 405] | 400.0 [305 to 404] | 400.0 [389 to 406] | 400.0 [386 to 400] | 400.0 [400 to 400] | 400.0 [378 to 404] | 400.0 [224 to 406] | 400.0 [300 to 401] | 400.0 [387 to 410] | 400.0 [400 to 400]

41. Secondary Outcome: Part 1, 2 and 3: Number of Participants With Anti-PDR001 Antibodies
Description: PDR001 immunogenicity was evaluated in serum samples. Patient anti-drug antibodies (ADA) status was defined as follows:
  * ADA-negative at baseline: ADA-negative sample at baseline
  * ADA-positive at baseline: ADA-positive sample at baseline
  * ADA-negative post-baseline: ADA-negative sample at baseline and at least 1 post-baseline sample, all of which are ADA-negative samples
  * Treatment-reduced ADA-positive: ADA-positive sample at baseline and at least 1 post-baseline sample, all of which are ADA-negative samples
  * Treatment-induced ADA-positive: ADA-negative sample at baseline and at least 1 treatment-induced ADA-positive sample
  * Treatment-boosted ADA-positive: ADA-positive sample at baseline and at least 1 treatment-boosted ADA-positive sample
  * ADA-inconclusive: patient who does not qualify for any of the above definitions or a patient for which the baseline sample is missing
Time Frame: Up to approximately 5 years
Population: All patients from Part 1, 2 and 3 who received at least 1 dose of NIR178 or PDR001 and had a determinant baseline immunogenicity (IG) sample and at least 1 determinant post-baseline IG sample for assessing anti-PDR001 antibodies. For the safety endpoints, patients at each study part with the same type of cancer who are treated at the same dose level and dosing schedule are pooled together, independently of the immune-oncology (IO) pretreatment status and RAS mutation status.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve + Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve + Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve + Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont
Number analyzed (Participants) | 11 | 23 | 12 | 13 | 24 | 11 | 52 | 27 | 13 | 10 | 6 | 13 | 21 | 19 | 17 | 6
Participants
  ADA-negative at baseline | 11 | 23 | 12 | 13 | 24 | 11 | 49 | 27 | 13 | 10 | 6 | 13 | 21 | 19 | 17 | 6
  ADA-positive at baseline | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA-negative post-baseline | 10 | 23 | 11 | 12 | 22 | 11 | 48 | 25 | 13 | 10 | 6 | 11 | 21 | 14 | 14 | 5
  Treatment-reduced ADA-positive | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-induced ADA-positive | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 5 | 3 | 1
  Treatment-boosted ADA-positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA-inconclusive | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Japan Safety Run-in: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications, which occurs within the first 28 days of treatment with NIR178 as single agent or in combination with PDR001 during the Japan safety run-in part of the study. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Time Frame: 28 days
Population: All patients in the Japan safety run-in who either met the minimum exposure criterion defined in the protocol and had sufficient safety evaluations, or had experienced a DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

43. Secondary Outcome: Japan Safety Run-in: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: as for outcome 36
Time Frame: Up to 0.7 years
Population: All patients from the Japan safety run-in who received at least 1 dose of NIR178 or PDR001.
Measure: Count of Participants; unit: Participants
Arm/Group | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Number analyzed (Participants) | 3 | 3 | 3
Participants
  AEs | 3 | 3 | 3
  Treatment-related AEs | 0 | 2 | 1
  SAEs | 2 | 1 | 1
  Treatment-related SAEs | 0 | 1 | 0
  Fatal SAEs | 0 | 0 | 0
  Treatment-related fatal SAEs | 0 | 0 | 0

44. Secondary Outcome: All Study Parts: Maximum Observed Plasma Concentration (Cmax) of NIR178
Description: Pharmacokinetic (PK) parameters were calculated based on NIR178 plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: Cycle 1 Day 1 (all), Cycle 1 Day 7 (1wk-on/1wk-off), Cycle 1 Day 14 (2wk-on/2wk-off) and Cycle 1 Day 28 (continuous dosing): pre-dose, 15 and 30 minutes, 1, 1.5, 2, 3, 4 and 8 hours after morning dose and 12 hours after evening dose. 1 cycle=28 days
Population: Patients in the pharmacokinetic analysis set (PAS) who received NIR178 and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one PK parameter and did not vomit within 4 hours after dosing with NIR178. Patients from the same ethnicity (Non-Japanese, Japanese) treated with the same formulation (capsule, tablet) at the same NIR178 dose level are pooled together.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- NIR178 160 mg Capsule in Non-Japanese (Part 1 and 2): Patients in Part 1 and 2 who received NIR178 160 mg as a capsule in combination with PDR001 400 mg every 4 weeks
- NIR178 240 mg Capsule in Non-Japanese (Part 1): Patients in Part 1 who received NIR178 240 mg as a capsule in combination with PDR001 400 mg every 4 weeks
- NIR178 160 mg Tablet in Non-Japanese (Part 3): Patients in Part 3 who received NIR178 160 mg as a film-coated tablet in combination with PDR001 400 mg every 4 weeks
Arm/Group | NIR178 160 mg Capsule in Non-Japanese (Part 1 and 2) | NIR178 240 mg Capsule in Non-Japanese (Part 1) | NIR178 160 mg Tablet in Non-Japanese (Part 3) | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Number analyzed (Participants) | 206 | 54 | 6 | 3 | 3 | 3
ng/mL
  Cycle 1 Day 1 (all regimens) | 129 (335.0) | 160 (247.8) | 75.1 (382.3) | 81.8 (99.9) | 30.1 (32.9) | 234 (70.9)
  Cycle 1 Day 7 (1 wk-on/1 wk-off): number analyzed (Participants) | 17 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 7 (1 wk-on/1 wk-off) | 576 (83.1) |  |  |  |  |
  Cycle 1 Day 14 (2 wk-on/2 wk-off): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 14 (2 wk-on/2 wk-off) | 392 (212.7) |  |  |  |  |
  Cycle 1 Day 28 (continuous): number analyzed (Participants) | 100 | 41 | 4 | 3 | 3 | 3
  Cycle 1 Day 28 (continuous) | 297 (291.4) | 622 (154.3) | 723 (295.5) | 311 (91.5) | 167 (40.9) | 3760 (39.6)

45. Secondary Outcome: All Study Parts: Time to Reach Maximum Plasma Concentration (Tmax) of NIR178
Description: Pharmacokinetic (PK) parameters were calculated based on NIR178 plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Median (Full Range); unit: hours
Arm/Group | NIR178 160 mg Capsule in Non-Japanese (Part 1 and 2) | NIR178 240 mg Capsule in Non-Japanese (Part 1) | NIR178 160 mg Tablet in Non-Japanese (Part 3) | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Number analyzed (Participants) | 206 | 54 | 6 | 3 | 3 | 3
hours
  Cycle 1 Day 1 (all regimens) | 2.00 [0.250 to 8.00] | 2.13 [0.50 to 8.00] | 1.50 [0.450 to 4.05] | 1.50 [1.47 to 1.50] | 1.50 [0.583 to 3.95] | 3.00 [2.03 to 3.03]
  Cycle 1 Day 7 (1 wk-on/1 wk-off): number analyzed (Participants) | 17 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 7 (1 wk-on/1 wk-off) | 1.45 [0.50 to 4.00] |  |  |  |  |
  Cycle 1 Day 14 (2 wk-on/2 wk-off): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 14 (2 wk-on/2 wk-off) | 1.97 [0.550 to 7.67] |  |  |  |  |
  Cycle 1 Day 28 (continuous): number analyzed (Participants) | 100 | 41 | 4 | 3 | 3 | 3
  Cycle 1 Day 28 (continuous) | 2.00 [0.267 to 8.00] | 2.02 [0.250 to 7.60] | 1.52 [0.50 to 3.00] | 1.43 [0.50 to 1.48] | 1.45 [0.50 to 1.50] | 2.87 [1.92 to 4.00]

46. Secondary Outcome: All Study Parts: Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours Post Dose (AUC0-12hr) of NIR178
Description: PK parameters were calculated based on NIR178 plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC0-12hr calculation.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | NIR178 160 mg Capsule in Non-Japanese (Part 1 and 2) | NIR178 240 mg Capsule in Non-Japanese (Part 1) | NIR178 160 mg Tablet in Non-Japanese (Part 3) | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Number analyzed (Participants) | 95 | 24 | 4 | 3 | 2 | 1
hr*ng/mL
  Cycle 1 Day 1 (all regimens) | 295 (198.3) | 487 (126.3) | 232 (437.4) | 170 (124.9) | 63.3 (88.0) | 550
  Cycle 1 Day 7 (1 wk-on/1 wk-off): number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 7 (1 wk-on/1 wk-off) | 1260 (63.2) |  |  |  |  |
  Cycle 1 Day 14 (2 wk-on/2 wk-off): number analyzed (Participants) | 7 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 14 (2 wk-on/2 wk-off) | 1680 (94.4) |  |  |  |  |
  Cycle 1 Day 28 (continuous): number analyzed (Participants) | 63 | 24 | 3 | 3 | 2 | 1
  Cycle 1 Day 28 (continuous) | 918 (187.5) | 1620 (147.9) | 938 (412.2) | 697 (131.8) | 242 (13.5) | 12800

47. Secondary Outcome: All Study Parts: Maximum Observed Plasma Concentration (Cmax) of NJI765 (NIR178 Metabolite)
Description: NJI765 is a NIR178 metabolite. PK parameters were calculated based on NJI765 plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | NIR178 160 mg Capsule in Non-Japanese (Part 1 and 2) | NIR178 240 mg Capsule in Non-Japanese (Part 1) | NIR178 160 mg Tablet in Non-Japanese (Part 3) | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Number analyzed (Participants) | 201 | 54 | 6 | 2 | 3 | 3
ng/mL
  Cycle 1 Day 1 (all regimens): number analyzed (Participants) | 201 | 54 | 6 | 0 | 3 | 3
  Cycle 1 Day 1 (all regimens) | 25.5 (85.2) | 33.7 (64.2) | 20.1 (99.2) |  | 25.9 (77.0) | 28.5 (99.9)
  Cycle 1 Day 7 (1 wk-on/1 wk-off): number analyzed (Participants) | 17 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 7 (1 wk-on/1 wk-off) | 62.9 (39.4) |  |  |  |  |
  Cycle 1 Day 14 (2 wk-on/2 wk-off): number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 14 (2 wk-on/2 wk-off) | 71.3 (43.3) |  |  |  |  |
  Cycle 1 Day 28 (continuous): number analyzed (Participants) | 96 | 40 | 4 | 2 | 3 | 3
  Cycle 1 Day 28 (continuous) | 42.6 (82.2) | 77.3 (49.9) | 54.1 (102.4) | 45.6 (74.0) | 53.9 (64.2) | 111 (36.6)

48. Secondary Outcome: All Study Parts: Time to Reach Maximum Plasma Concentration (Tmax) of NJI765 (NIR178 Metabolite)
Description: NJI765 is a NIR178 metabolite. Pharmacokinetic (PK) parameters were calculated based on NJI765 plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Median (Full Range); unit: hours
Arm/Group | NIR178 160 mg Capsule in Non-Japanese (Part 1 and 2) | NIR178 240 mg Capsule in Non-Japanese (Part 1) | NIR178 160 mg Tablet in Non-Japanese (Part 3) | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Number analyzed (Participants) | 201 | 54 | 6 | 2 | 3 | 3
hours
  Cycle 1 Day 1 (all regimens): number analyzed (Participants) | 201 | 54 | 6 | 0 | 3 | 3
  Cycle 1 Day 1 (all regimens) | 2.00 [0.250 to 8.05] | 2.08 [0.50 to 8.00] | 2.10 [0.450 to 4.05] |  | 1.95 [0.583 to 2.00] | 3.00 [2.03 to 3.03]
  Cycle 1 Day 7 (1 wk-on/1 wk-off): number analyzed (Participants) | 17 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 7 (1 wk-on/1 wk-off) | 1.50 [0.50 to 4.00] |  |  |  |  |
  Cycle 1 Day 14 (2 wk-on/2 wk-off): number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 14 (2 wk-on/2 wk-off) | 1.98 [0.550 to 3.00] |  |  |  |  |
  Cycle 1 Day 28 (continuous): number analyzed (Participants) | 96 | 40 | 4 | 2 | 3 | 3
  Cycle 1 Day 28 (continuous) | 2.00 [0.483 to 8.03] | 2.10 [0.250 to 7.88] | 0.750 [0.50 to 2.03] | 2.23 [1.43 to 3.02] | 1.45 [0.50 to 1.50] | 2.87 [1.92 to 4.00]

49. Secondary Outcome: All Study Parts: Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours Post Dose (AUC0-12hr) of NJI765 (NIR178 Metabolite)
Description: NJI765 is a NIR178 metabolite. PK parameters were calculated based on NJI765 plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC0-12hr calculation.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | NIR178 160 mg Capsule in Non-Japanese (Part 1 and 2) | NIR178 240 mg Capsule in Non-Japanese (Part 1) | NIR178 160 mg Tablet in Non-Japanese (Part 3) | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Number analyzed (Participants) | 62 | 20 | 2 | 0 | 3 | 1
hr*ng/mL
  Cycle 1 Day 1 (all regimens) | 98.2 (87.1) | 122 (75.6) | 77.1 (35.9) |  | 117 (68.2) | 119
  Cycle 1 Day 7 (1 wk-on/1 wk-off): number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 7 (1 wk-on/1 wk-off) | 243 (57.5) |  |  |  |  |
  Cycle 1 Day 14 (2 wk-on/2 wk-off): number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 14 (2 wk-on/2 wk-off) | 288 (23.7) |  |  |  |  |
  Cycle 1 Day 28 (continuous): number analyzed (Participants) | 41 | 16 | 2 | 0 | 2 | 1
  Cycle 1 Day 28 (continuous) | 214 (76.6) | 382 (43.7) | 226 (147.0) |  | 277 (69.0) | 362

50. Secondary Outcome: All Study Parts: Maximum Observed Serum Concentration (Cmax) of PDR001
Description: PK parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: First dose (Cycle 1 Day 1 or Cycle 2 Day 1 for Japanese patients treated with NIR178 80 or 160 mg) and Cycle 3 Day 1: pre-infusion, 1, 168, 336, 504 and 672 hours after end of infusion. Average duration of infusion=30 minutes. 1 cycle=28 days
Population: Patients in the pharmacokinetic analysis set (PAS) who received PDR001 and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one PK parameter and did not vomit within 4 hours after dosing with NIR178. Patients from the same ethnicity (Non-Japanese, Japanese) treated at the same PDR001 dose level are pooled together.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Non-Japanese Patients: Patients in Parts 1, 2 and 3 who received NIR178 (any dose level) in combination with PDR001 400 mg every 4 weeks
- Japanese Patients: Patients in the Japanese safety run-in part who received NIR178 (any dose level) in combination with PDR001 400 mg every 4 weeks
Arm/Group | Non-Japanese Patients | Japanese Patients
Number analyzed (Participants) | 257 | 3
µg/mL
  First dose (Cycle 1 Day 1 or Cycle 2 Day 1) | 93.2 (30.8) | 85.0 (12.8)
  Cycle 3 Day 1: number analyzed (Participants) | 132 | 1
  Cycle 3 Day 1 | 126 (37.4) | 119

51. Secondary Outcome: All Study Parts: Time to Reach Maximum Serum Concentration (Tmax) of PDR001
Description: PK parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 50
Population: as for outcome 50
Measure: Median (Full Range); unit: hours
Arm/Group | Non-Japanese Patients | Japanese Patients
Number analyzed (Participants) | 257 | 3
hours
  First dose (Cycle 1 Day 1 or Cycle 2 Day 1) | 1.50 [0.333 to 718] | 1.50 [1.48 to 1.52]
  Cycle 3 Day 1: number analyzed (Participants) | 132 | 1
  Cycle 3 Day 1 | 1.50 [0.550 to 358] | 1.65 [1.65 to 1.65]

52. Secondary Outcome: All Study Parts: Area Under the Serum Concentration-time Curve From Time Zero to 28 Days Post Dose (AUC0-28day) of PDR001
Description: PK parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC0-28day calculation.
Time Frame: as for outcome 50
Population: as for outcome 50
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/mL
Arm/Group | Non-Japanese Patients | Japanese Patients
Number analyzed (Participants) | 236 | 3
day*µg/mL
  First dose (Cycle 1 Day 1 or Cycle 2 Day 1) | 1140 (31.2) | 1110 (13.9)
  Cycle 3 Day 1: number analyzed (Participants) | 36 | 0
  Cycle 3 Day 1 | 2030 (41.3) |

53. Post Hoc Outcome: All-Collected Deaths
Description: On-treatment and post-treatment safety follow-up deaths were collected from first dose of study medication to 150 days after last dose of NIR178+PDR001. Survival follow-up deaths were collected from 151 days after last dose of NIR178+PDR001 until end of study. All deaths refer to the sum of on-treatment and post-treatment safety follow-up deaths plus survival follow-up deaths.
Time Frame: On-treatment and safety follow-up (FU) deaths: up to 4.3 years (Part 1), 5.1 years (Part 2), 0.9 years (Part 3) and 0.9 years (JSR). Survival FU deaths: up to 4.3 years (Part 1), 5.1 years (Part 2) and 0.9 years (Part 3) and 0.9 years (JSR)
Population: All patients who received at least one dose of study treatment. Patients at each study part with the same type of cancer who are treated at the same dose level and dosing schedule are pooled together, independently of the immune-oncology (IO) pretreatment status and RAS mutation status.
Measure: Number; unit: participants
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve + Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve + Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve + Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont
Number analyzed (Participants) | 11 | 23 | 14 | 14 | 26 | 12 | 58 | 30 | 16 | 13 | 6 | 15 | 22 | 20 | 20 | 6 | 3 | 3 | 3
participants
  On-treatment and post-treatment safety follow-up deaths | 4 | 6 | 10 | 6 | 8 | 4 | 22 | 9 | 7 | 9 | 2 | 2 | 6 | 4 | 6 | 4 | 2 | 0 | 1
  Survival follow-up deaths: number analyzed (Participants) | 7 | 17 | 4 | 8 | 18 | 8 | 36 | 21 | 9 | 4 | 4 | 13 | 16 | 16 | 14 | 2 | 0 | 0 | 1
  Survival follow-up deaths | 3 | 7 | 3 | 4 | 12 | 4 | 22 | 12 | 8 | 2 | 3 | 7 | 8 | 9 | 7 | 1 |  |  | 1
  All deaths | 7 | 13 | 13 | 10 | 20 | 8 | 44 | 21 | 15 | 11 | 5 | 9 | 14 | 13 | 13 | 5 | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: On-treatment and post-treatment safety follow-up: from first dose of study treatment to 150 days after last dose of NIR178+PDR001, up to 4.3 years (Part 1), 5.1 years (Part 2), 0.9 years (Part 3) and 0.9 years (Japan safety run-in; JSR). Deaths in survival period: from 151 days after last dose of NIR178+PDR001 until end of study, up to 4.3 years (Part 1), 5.1 years (Part 2), 0.9 years (Part 3) and 0.9 years (JSR).
Description: Deaths in the survival period are not considered Adverse Events (AEs). No AEs were collected in the survival period.
Groups:
- Part 1: RCC naïve 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with renal cell carcinoma (RCC) who had not been previously treated with immuno-oncology therapy. Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: RCC naïve + Pre 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with renal cell carcinoma (RCC), naïve and pretreated with immuno-oncology therapy. Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: Pancreatic 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with pancreatic cancer. Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: Urothelial 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with urothelial cancer. Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: H-N naïve + Pre 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with squamous cell carcinoma of head and neck (HNSCC), naïve and pretreated with immuno-oncology therapy. Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: H-N Pre 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with squamous cell carcinoma of head and neck (HNSCC) who had been pretreated with immuno-oncology therapy. Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: MSS CRC 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with microsatellite stable colorectal cancer (MSS CRC) and RAS wildtype, RAS mutant and RAS unknown status. Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: TNBC 160 mg; Part 3: TNBC 160 mg Cont: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with triple negative breast cancer (TNBC). Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: Melanoma naïve + Pre 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with cutaneous melanoma, naïve and pretreated with immuno-oncology therapy. Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: DLBCL 160 mg: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with diffuse large B-cell lymphoma (DLBCL). Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: DLBCL 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with diffuse large B-cell lymphoma (DLBCL). Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: mCRPC 240 mg: NIR178 240 mg twice daily continuous in combination with PDR001 in patients with metastatic castration resistant prostate cancer (mCRPC). Safety data up to 150 days after last dose of NIR178+PDR001
- Part 2: NSCLC 160 mg Cont: NIR178 160 mg twice daily continuous in combination with PDR001 in patients with non-small cell lung cancer (NSCLC). Safety data up to 150 days after last dose of NIR178+PDR001
- Part 2: NSCLC 160 mg 2wk-on/2wk-off: NIR178 160 mg twice daily 2 weeks on/2 weeks off in combination with PDR001 in patients with non-small cell lung cancer (NSCLC). Safety data up to 150 days after last dose of NIR178+PDR001
- Part 2: NSCLC 160 mg 1wk-on/1wk-off: NIR178 160 mg twice daily 1 week on/1 week off in combination with PDR001 in patients with non-small cell lung cancer (NSCLC). Safety data up to 150 days after last dose of NIR178+PDR001
- JSR: 80 mg Cont: NIR178 80 mg twice daily continuous in combination with PDR001 (starting Cycle 2 Day 1) in the Japan safety run-in. Safety data up to 150 days after last dose of NIR178+PDR001
- JSR: 160 mg Cont: NIR178 160 mg twice daily continuous in combination with PDR001 (starting Cycle 2 Day 1) in the Japan safety run-in. Safety data up to 150 days after last dose of NIR178+PDR001
- JSR: 240 mg Cont: NIR178 140 mg twice daily continuous in combination with PDR001 (starting Cycle 1 Day 1) in the Japan safety run-in. Safety data up to 150 days after last dose of NIR178+PDR001
- Part 1: RCC naïve 160 mg_Survival Period; Part 1: RCC naïve + Pre 240 mg_Survival Period; Part 1: Pancreatic 160 mg_Survival Period; Part 1: Urothelial 160 mg_Survival Period; Part 1: H-N naïve + Pre 160 mg_Survival Period; Part 1: H-N Pre 240 mg_Survival Period; Part 1: MSS CRC 160 mg_Survival Period; Part 1: TNBC 160 mg_Survival Period; Part 1: Melanoma naïve + Pre 160 mg_Survival Period; Part 1: DLBCL 160 mg_Survival Period; Part 1: DLBCL 240 mg_Survival Period; Part 1: mCRPC 240 mg_Survival Period; Part 2: NSCLC 160 mg cont_Survival Period; Part 2: NSCLC 160 mg 2wk-on/2wk-off_Survival Period; Part 2: NSCLC 160 mg 1wk-on/1wk-off_Survival Period; Part 3: TNBC 160 mg cont_Survival Period; JSR: 80 mg cont_Survival Period; JSR: 160 mg cont_Survival Period; JSR: 240 mg cont_Survival Period: Deaths collected in the survival follow-up period (starting from Day 151 after last dose of NIR178+PDR001). No AEs were collected during this period.
Arm/Group | Part 1: RCC naïve 160 mg | Part 1: RCC naïve + Pre 240 mg | Part 1: Pancreatic 160 mg | Part 1: Urothelial 160 mg | Part 1: H-N naïve + Pre 160 mg | Part 1: H-N Pre 240 mg | Part 1: MSS CRC 160 mg | Part 1: TNBC 160 mg | Part 1: Melanoma naïve + Pre 160 mg | Part 1: DLBCL 160 mg | Part 1: DLBCL 240 mg | Part 1: mCRPC 240 mg | Part 2: NSCLC 160 mg Cont | Part 2: NSCLC 160 mg 2wk-on/2wk-off | Part 2: NSCLC 160 mg 1wk-on/1wk-off | Part 3: TNBC 160 mg Cont | JSR: 80 mg Cont | JSR: 160 mg Cont | JSR: 240 mg Cont | Part 1: RCC naïve 160 mg_Survival Period | Part 1: RCC naïve + Pre 240 mg_Survival Period | Part 1: Pancreatic 160 mg_Survival Period | Part 1: Urothelial 160 mg_Survival Period | Part 1: H-N naïve + Pre 160 mg_Survival Period | Part 1: H-N Pre 240 mg_Survival Period | Part 1: MSS CRC 160 mg_Survival Period | Part 1: TNBC 160 mg_Survival Period | Part 1: Melanoma naïve + Pre 160 mg_Survival Period | Part 1: DLBCL 160 mg_Survival Period | Part 1: DLBCL 240 mg_Survival Period | Part 1: mCRPC 240 mg_Survival Period | Part 2: NSCLC 160 mg cont_Survival Period | Part 2: NSCLC 160 mg 2wk-on/2wk-off_Survival Period | Part 2: NSCLC 160 mg 1wk-on/1wk-off_Survival Period | Part 3: TNBC 160 mg cont_Survival Period | JSR: 80 mg cont_Survival Period | JSR: 160 mg cont_Survival Period | JSR: 240 mg cont_Survival Period
All-Cause Mortality (participants affected / at risk) | 4/11 | 6/23 | 10/14 | 6/14 | 8/26 | 4/12 | 22/58 | 9/30 | 7/16 | 9/13 | 2/6 | 2/15 | 6/22 | 4/20 | 6/20 | 4/6 | 2/3 | 0/3 | 1/3 | 3/7 | 7/17 | 3/4 | 4/8 | 12/18 | 4/8 | 22/36 | 12/21 | 8/9 | 2/4 | 3/4 | 7/13 | 8/16 | 9/16 | 7/14 | 1/2 | 0/0 | 0/0 | 1/1
Serious Adverse Events (participants affected / at risk) | 3/11 | 7/23 | 9/14 | 7/14 | 16/26 | 5/12 | 28/58 | 14/30 | 4/16 | 7/13 | 0/6 | 5/15 | 11/22 | 9/20 | 7/20 | 3/6 | 2/3 | 1/3 | 1/3 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 10/11 | 22/23 | 14/14 | 14/14 | 25/26 | 12/12 | 52/58 | 29/30 | 14/16 | 13/13 | 5/6 | 14/15 | 22/22 | 16/20 | 17/20 | 6/6 | 3/3 | 2/3 | 3/3 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: RCC naïve 160 mg (N=11) | Part 1: RCC naïve + Pre 240 mg (N=23) | Part 1: Pancreatic 160 mg (N=14) | Part 1: Urothelial 160 mg (N=14) | Part 1: H-N naïve + Pre 160 mg (N=26) | Part 1: H-N Pre 240 mg (N=12) | Part 1: MSS CRC 160 mg (N=58) | Part 1: TNBC 160 mg (N=30) | Part 1: Melanoma naïve + Pre 160 mg (N=16) | Part 1: DLBCL 160 mg (N=13) | Part 1: DLBCL 240 mg (N=6) | Part 1: mCRPC 240 mg (N=15) | Part 2: NSCLC 160 mg Cont (N=22) | Part 2: NSCLC 160 mg 2wk-on/2wk-off (N=20) | Part 2: NSCLC 160 mg 1wk-on/1wk-off (N=20) | Part 3: TNBC 160 mg Cont (N=6) | JSR: 80 mg Cont (N=3) | JSR: 160 mg Cont (N=3) | JSR: 240 mg Cont (N=3) | Part 1: RCC naïve 160 mg_Survival Period (N=0) | Part 1: RCC naïve + Pre 240 mg_Survival Period (N=0) | Part 1: Pancreatic 160 mg_Survival Period (N=0) | Part 1: Urothelial 160 mg_Survival Period (N=0) | Part 1: H-N naïve + Pre 160 mg_Survival Period (N=0) | Part 1: H-N Pre 240 mg_Survival Period (N=0) | Part 1: MSS CRC 160 mg_Survival Period (N=0) | Part 1: TNBC 160 mg_Survival Period (N=0) | Part 1: Melanoma naïve + Pre 160 mg_Survival Period (N=0) | Part 1: DLBCL 160 mg_Survival Period (N=0) | Part 1: DLBCL 240 mg_Survival Period (N=0) | Part 1: mCRPC 240 mg_Survival Period (N=0) | Part 2: NSCLC 160 mg cont_Survival Period (N=0) | Part 2: NSCLC 160 mg 2wk-on/2wk-off_Survival Period (N=0) | Part 2: NSCLC 160 mg 1wk-on/1wk-off_Survival Period (N=0) | Part 3: TNBC 160 mg cont_Survival Period (N=0) | JSR: 80 mg cont_Survival Period (N=0) | JSR: 160 mg cont_Survival Period (N=0) | JSR: 240 mg cont_Survival Period (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Autoimmune myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gaze palsy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
General physical health deterioration (General disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Large intestine infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Scrotal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urogenital infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary tumour thrombotic microangiopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peyronie's disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: RCC naïve 160 mg (N=11) | Part 1: RCC naïve + Pre 240 mg (N=23) | Part 1: Pancreatic 160 mg (N=14) | Part 1: Urothelial 160 mg (N=14) | Part 1: H-N naïve + Pre 160 mg (N=26) | Part 1: H-N Pre 240 mg (N=12) | Part 1: MSS CRC 160 mg (N=58) | Part 1: TNBC 160 mg (N=30) | Part 1: Melanoma naïve + Pre 160 mg (N=16) | Part 1: DLBCL 160 mg (N=13) | Part 1: DLBCL 240 mg (N=6) | Part 1: mCRPC 240 mg (N=15) | Part 2: NSCLC 160 mg Cont (N=22) | Part 2: NSCLC 160 mg 2wk-on/2wk-off (N=20) | Part 2: NSCLC 160 mg 1wk-on/1wk-off (N=20) | Part 3: TNBC 160 mg Cont (N=6) | JSR: 80 mg Cont (N=3) | JSR: 160 mg Cont (N=3) | JSR: 240 mg Cont (N=3) | Part 1: RCC naïve 160 mg_Survival Period (N=0) | Part 1: RCC naïve + Pre 240 mg_Survival Period (N=0) | Part 1: Pancreatic 160 mg_Survival Period (N=0) | Part 1: Urothelial 160 mg_Survival Period (N=0) | Part 1: H-N naïve + Pre 160 mg_Survival Period (N=0) | Part 1: H-N Pre 240 mg_Survival Period (N=0) | Part 1: MSS CRC 160 mg_Survival Period (N=0) | Part 1: TNBC 160 mg_Survival Period (N=0) | Part 1: Melanoma naïve + Pre 160 mg_Survival Period (N=0) | Part 1: DLBCL 160 mg_Survival Period (N=0) | Part 1: DLBCL 240 mg_Survival Period (N=0) | Part 1: mCRPC 240 mg_Survival Period (N=0) | Part 2: NSCLC 160 mg cont_Survival Period (N=0) | Part 2: NSCLC 160 mg 2wk-on/2wk-off_Survival Period (N=0) | Part 2: NSCLC 160 mg 1wk-on/1wk-off_Survival Period (N=0) | Part 3: TNBC 160 mg cont_Survival Period (N=0) | JSR: 80 mg cont_Survival Period (N=0) | JSR: 160 mg cont_Survival Period (N=0) | JSR: 240 mg cont_Survival Period (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 5 | 5 | 0 | 5 | 4 | 3 | 3 | 1 | 2 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 5 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 4 | 1 | 3 | 0 | 9 | 2 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 6 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 7 | 1 | 2 | 4 | 1 | 9 | 2 | 1 | 3 | 1 | 2 | 8 | 3 | 8 | 2 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 | 8 | 0 | 4 | 4 | 1 | 12 | 3 | 0 | 1 | 0 | 3 | 4 | 1 | 2 | 3 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 5 | 1 | 5 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 1 | 5 | 4 | 5 | 6 | 2 | 13 | 9 | 4 | 2 | 0 | 5 | 5 | 3 | 3 | 4 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 3 | 4 | 0 | 12 | 5 | 0 | 2 | 0 | 0 | 5 | 3 | 4 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Administration site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Asthenia (General disorders) | 2 | 5 | 1 | 2 | 0 | 0 | 3 | 5 | 4 | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Catheter site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chills (General disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 4 | 5 | 5 | 2 | 11 | 3 | 20 | 10 | 3 | 1 | 0 | 4 | 11 | 6 | 5 | 3 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Feeling of body temperature change (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 2 | 2 | 2 | 3 | 2 | 0 | 5 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 1 | 2 | 1 | 4 | 4 | 0 | 9 | 9 | 0 | 4 | 1 | 2 | 2 | 4 | 1 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 2 | 1 | 2 | 1 | 0 | 0 | 5 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urogenital infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0 | 2 | 3 | 1 | 11 | 9 | 1 | 0 | 1 | 3 | 2 | 4 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Amylase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 4 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 1 | 2 | 3 | 1 | 14 | 9 | 1 | 1 | 0 | 3 | 2 | 4 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 1 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Human chorionic gonadotropin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 0 | 0 | 4 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
SARS-CoV-2 test negative (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 7 | 5 | 6 | 0 | 17 | 4 | 2 | 3 | 0 | 2 | 6 | 5 | 3 | 1 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 1 | 0 | 4 | 3 | 0 | 3 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 0 | 4 | 0 | 9 | 8 | 0 | 0 | 0 | 2 | 3 | 3 | 1 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1 | 3 | 2 | 0 | 5 | 4 | 1 | 0 | 1 | 3 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 4 | 4 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 2 | 5 | 2 | 1 | 1 | 1 | 4 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 1 | 2 | 3 | 4 | 1 | 1 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 0 | 3 | 2 | 2 | 1 | 0 | 4 | 1 | 0 | 2 | 0 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Panic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Leukocyturia (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peyronie's disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 4 | 4 | 0 | 11 | 10 | 1 | 2 | 0 | 2 | 6 | 2 | 3 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4 | 2 | 1 | 8 | 6 | 1 | 2 | 0 | 1 | 5 | 1 | 5 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1 | 2 | 1 | 8 | 3 | 2 | 1 | 0 | 1 | 5 | 2 | 3 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 2 | 5 | 0 | 2 | 3 | 1 | 3 | 1 | 1 | 2 | 0 | 4 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Angiopathy (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Flushing (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hot flush (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03207867/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03207867/SAP_001.pdf